CLINICAL TRIAL: NCT02165956
Title: Effect of a New Food Product on Weight Gain During First Infancy
Brief Title: Effect of a New Infant Cereal on Weight Gain
Acronym: CEOBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorios Ordesa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CEOBE-01-011
Record Dates: First submitted 2014-06-11; First posted 2014-06-18 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Infant Development
Keywords: Cereals; Obesity; Complementary Feeding
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Infant Cereal (Experimental): The amount of cereal administered will be free and from 6 to 12 months of age.
  Interventions: Dietary Supplement: New Infant Cereal
- Standard Infant Cereal (Active Comparator): The amount of cereal administered will be free and from 6 to 12 months of age.
  Interventions: Dietary Supplement: Standard Infant Cereal

INTERVENTIONS:
Dietary Supplement: New Infant Cereal — New Infant Cereal
  Arms: New Infant Cereal
Dietary Supplement: Standard Infant Cereal — Standard Infant Cereal
  Arms: Standard Infant Cereal

SUMMARY:
The purpose of this study is to determine whether a new infant cereal has an effect on weight gain and intestinal microbiota compared to a standard cereal in healthy infants .

DETAILED DESCRIPTION:
This is a multicenter, controlled, randomized, prospective, parallel-group, double-blind study to evaluate the effect of a new infant cereal supplemented with prebiotics, probiotics, vegetable proteins and a special blend of starches on weight gain and intestinal microbiota in healthy infants from 6 to 12 moths of age. Patients will be randomized to receive either the new infant cereal or a standard cereal.

ELIGIBILITY:
Inclusion Criteria:

* Lactating babies
* 6 months of age
* Informed consent signed by parents

Exclusion Criteria:

* Malformations, diseases or conditions that may alter development and/or nutritional status
* Born very and extremely preterm (<32 weeks of gestational age)

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Changes in nutritional status | At 6, 9, 12, 15 and 18 months of age
  Difference between groups measured by a composite of nutritional parameters(weight, height, perimeters and skin fold measurements).

SECONDARY OUTCOMES:
Changes in appetite | At 6, 9, 12, 15 and 18 months of age
  Differences between groups measured by a 3-day food record.
Tolerability of study product | At 6, 9, 12, 15 and 18 months of age
  Differences between groups measured by frequency and type of a composite of gastrointestinal symptoms (regurgitation, irritability, flatulence and crying).
Changes in intestinal microbiota | At 6, 9, 12 and 18 months of age
  Differences between groups measured by the analysis of faecal samples.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Alberto Moreno, Professor, Principal Investigator — Universidad de Zaragoza; Gerardo Rodríguez, Professor, Principal Investigator — Universidad de Zaragoza; Mª Luisa Álvarez, Principal Investigator — Universidad de Zaragoza; Mª Jesús Cabero, Principal Investigator — University of Cantabria; Laura Monje, Principal Investigator — University of Cantabria
Locations (5):
- Spain (5):
  - Consultorio de Soto de la Marina, Soto de la Marina, Cantabria
  - Centro de Salud Santo Grial, Huesca
  - Centro de Salud Perpetuo Socorro, Huesca
  - Centro de Salud Isabel II-Centro, Santander
  - Centro de Salud El Alisal, Santander

REFERENCES:
- [Result] Rodríguez G, Cabero MJ, Samper P, Álvarez ML, Monje L, Morera M, Rivero M, García-Fuentes M, Moreno L. Complementary feeding and infant body composition in northern Spain. Ann Nutr Metab. 2013;63 (suppl 1):1-1960. PO908.
- [Result] Rodriguez G, Cabero MJ, Morera M, Samper P, Álvarez ML, Monje L, Moreno L, García-Fuentes M, Rivero M. Intake pattern of infant complementary feeding in two populations in Northern Spain. JPGN. 2013;56(Suppl 2):486. PO-N-0283.
- [Result] Morera M, Rodríguez G, Cabero MJ, Samper P, Álvarez ML, Monje L, Miralles A, Álvarez L, Rivero M, García-Fuentes M, Moreno L. Rapid weight gain during complementary feeding period and overweight risk. JPGN. 2014;58(Suppl 1):456. PO-N-0274.